CLINICAL TRIAL: NCT04242407
Title: A Double-Blind, Placebo-Controlled Evaluation of the Dexmedetomidine Transdermal System for Postoperative Analgesia Following Abdominoplasty
Brief Title: Evaluating Efficacy of the Dexmedetomidine Transdermal System for Postoperative Analgesia Following Abdominoplasty
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Teikoku Pharma USA, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TPU-DMT-02-1908
Record Dates: First submitted 2020-01-22; First posted 2020-01-27 (Actual); Last update posted 2020-07-23 (Actual); Status verified 2020-07

CONDITIONS: Pain, Postoperative
Keywords: Abdominoplasty; Pain; Dexmedetomidine; Transdermal; Postoperative; DMTS
MeSH Terms: conditions — Pain, Postoperative; Pain

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized in 1:1 ratio to receive DMTS or matching placebo.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The sponsor, the investigator, personnel at the clinical study unit who are directly involved with monitoring and/or performing study procedures and assessments, and the subjects will be blinded to treatment assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- DMTS (Active Comparator): DMTS applied to the upper arm
  Interventions: Drug: DMTS
- Placebo (Placebo Comparator): Placebo system (with no drug) to match DMTS applied to the upper arm
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: DMTS — DMTS applied before surgery and worn for 96 hours
  Arms: DMTS
Drug: Placebo — Matching patches that have no active drug applied before surgery and worn for 96 hours
  Arms: Placebo

SUMMARY:
The primary objective of this study is to evaluate the analgesic efficacy of Dexmedetomidine Transdermal System (DMTS), compared with placebo, in participants following abdominoplasty.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, one-time application study of DMTS or matching placebo over a 4-day treatment period.

Eligible subjects will be randomized in 1:1 ratio to receive DMTS or matching placebo. Subjects will reside at the clinical study unit for up to a total of 7 days. The surgical procedure, the intraoperative anesthesia, and the medication used for infiltration of the wound for local anesthesia before the last stitch will be standardized. During the postoperative period in the clinical study unit, recovery procedures will be standardized.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily provide written informed consent.
2. Male or female, ≥ 18 years of age.
3. Scheduled to undergo a full abdominoplasty (including repair of small incidental abdominal hernias but not including liposuction).
4. Have a physical status classification of 1 or 2 per the American Society of Anesthesiology.
5. Female subjects are eligible only if all the following apply:

   1. Not pregnant, not lactating, and not planning to become pregnant during the study or for 1 menstrual cycle thereafter
   2. Surgically sterile; or at least 2 years postmenopausal; or have a monogamous partner who is surgically sterile; or have a same gender sex partner; or is using double-barrier contraception; or practicing abstinence; or using an insertable, injectable, transdermal, or combination oral contraceptive for 3 months prior to the study, during the study, and for 1 month following the study
6. Male subjects with female sex partners of childbearing potential must be surgically sterile or commit to use a reliable method of birth control during the study and for 1 month following the study.
7. Have a body weight > 58 kg and a BMI of 20 to 38 kg/m2, inclusive.
8. Able to understand the study procedures, comply with all study procedures, and agree to participate in the study program for its full duration.

Exclusion Criteria:

1. Known sensitivity to dexmedetomidine or any excipient in the DMTS/placebo or to any peri- or postoperative medication whose use is required in this study.
2. Skin abnormality (eg, scar, tattoo) or unhealthy skin condition (eg, burns, wounds) at the DMTS/matching placebo system application site, according to examination by the investigator at screening or admission to the clinic prior to surgery.
3. Clinically significant abnormal clinical laboratory test value.
4. History of deep vein thrombosis or factor V Leiden deficiency.
5. History of or positive test results for the human immunodeficiency virus (HIV), hepatitis B, or hepatitis C.
6. History or clinical manifestations of: a significant renal, hepatic, cardiovascular, metabolic, neurologic, or psychiatric condition; congestive heart failure, peptic ulcer, gastrointestinal bleeding, or other condition that may preclude participation in the study.
7. History of physician-diagnosed migraine, frequent non-vascular headaches (> 5 per month), seizures, or are currently taking anticonvulsants.
8. Have another painful physical condition that may confound the assessments of postoperative pain.
9. History of syncope or other syncopal attacks.
10. Present and/or significant history of postural hypotension (determined through examination by the investigator or designee), or history of severe dizziness or fainting on standing in the opinion of the investigator.
11. Evidence of a clinically significant 12-lead ECG abnormality.
12. Supine heart rate < 60 or > 100 bpm, systolic blood pressure (BP) < 90 or > 140 mmHg, or diastolic BP < 60 or > 90 mmHg, when measured in triplicate: after being supine for at least 5 minutes; after sitting for at least 2 minutes; and after standing for at least 2 minutes.
13. History of alcohol abuse or prescription/illicit drug abuse within the previous 5 years.
14. Positive results on the urine drug screen or alcohol breath test indicative of drugs of abuse or alcohol use at screening and/or clinic check-in.
15. Receiving or have received opioid therapy chronically for > 2 weeks within the month prior to dosing of the study drug.
16. Receiving concurrent therapy that can interfere with the evaluation of efficacy or safety, such as any drug that in the investigator's opinion may exert significant analgesic properties or act synergistically with dexmedetomidine.
17. Used of any natural health products (including chaparral, comfrey, germander, jin bu huan, kava, pennyroyal, skullcap, St. John's wort, or valerian, and excluding vitamins or mineral supplements) within 14 days prior to study drug administration and throughout the study, unless in the opinion of the investigator or designee, the product will not interfere with the study procedures or data integrity, or compromise the safety of the subject.
18. Had symptoms of an upper respiratory tract infection within 14 days prior to dosing of the study drug.
19. Utilized oral or injectable corticosteroids within 14 days prior to dosing of the study drug (intranasal and topical corticosteroid use during this time period is allowed).
20. Received any investigational product within 30 days prior to dosing of the study drug.
21. Received DMTS in a previous clinical trial.
22. Sensitivity to opioids, nonsteroidal anti-inflammatory drugs, or antibiotics.
23. In the opinion of the investigator or designee, is considered unsuitable for study entry and/or is unlikely to comply with the study protocol for any reason.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Estimated)
Dates: Start 2020-07-07 (Actual); Primary Completion 2021-02-01 (Estimated); Study Completion 2021-02-01 (Estimated)

PRIMARY OUTCOMES:
Time-interval weighted summed pain intensity (SPI) with activity | 4 to 96 hours following surgery
  The SPI measured using the 11-point (0 to 10) numeric rating scale, where 0 is equal to no pain and 10 is equal to worst pain, with activity (ie, splinted cough with pillow).

SECONDARY OUTCOMES:
Time-interval weighted summed pain intensity (SPI) (rest and activity) | 4 to 96 hours following surgery
  The SPI measured using the 11-point (0 to 10) numeric rating scale, where 0 is equal to no pain and 10 is equal to worst pain, measured at rest and with activity over various time intervals
Rescue Medication | 4 to 96 hours following surgery
  The proportion of subjects using rescue analgesic medication
Rescue Medication time | 4 to 96 hours following surgery
  The time to first use of rescue analgesic medication
Rescue Medication units | 4 to 96 hours following surgery
  Total dose of rescue analgesic medication (in morphine-equivalent units)
Integrated Pain score and Rescue Medication | 4 to 96 hours following surgery
  Integrated assessments of summed pain intensity (SPI) using the 11-point (0 to 10) numeric rating scale, where 0 is equal to no pain and 10 is equal to worst pain, measured at the time Rescue Medication was administered.

CONTACTS AND LOCATIONS:
Overall Officials: James Song, MS, MBA, Study Director — Teikoku Pharma USA, Inc.
Locations (4):
- United States (4):
  - Arizona Research Center, Phoenix, Arizona
  - HD Research, Bellaire, Texas
  - Endeavor Clinical Trials, San Antonio, Texas
  - JBR Clinical Research, Salt Lake City, Utah